CLINICAL TRIAL: NCT05674968
Title: A Pilot Feasibility Randomized Control Trial of the Managing Challenging Behaviors in ADHD
Brief Title: Managing Challenging Behaviors-ADHD
Acronym: MCB-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, James T. Craig, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY02001611
Record Dates: First submitted 2022-12-19; First posted 2023-01-09 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: 60 families will be enrolled in the study. The researchers will use block randomization to assign half to the treatment group and half to a wait-list control group. Participants will be blocked by gender and condition.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Managing Challenging Behaviors in ADHD (Experimental): This is a 7-session behavioral parent training delivered to children ages 3-7 referred to the study after an initial ADHD diagnosis or when challenging behaviors are identified by their medical provider.
  Interventions: Behavioral: Managing Challenging Behaviors in ADHD; Psychosocial program
- Wait List (No Intervention): Families assigned to the wait list will complete measures at baseline, 14 weeks, and 24 weeks. After 24 weeks they will be offered the experimental treatment.

INTERVENTIONS:
Behavioral: Managing Challenging Behaviors in ADHD; Psychosocial program — MCB-ADHD is a brief Behavioral Parent Training (BPT) program delivered to caregivers and children together. THe researchers have specially designed this program to be flexible so that it can be delivered over telehealth and/or in-person. All sessions are guided by web-based tool to provide parent support materials and direct the work to be completed in session. MCB-ADHD combines brief BPT skills modules adapted from an established evidence-based BPT called Helping the Noncompliant Child (HNC; McMahon & Forehand, 2003) with high quality psychoeducation and advocacy training that were developed by the investigators specifically for use in this project. Families receive 4 sessions adapted from HNC focused on behavior management and 2 sessions focused on education and empowerment.
  Arms: Managing Challenging Behaviors in ADHD

SUMMARY:
The purpose of this study is to test whether short, time-limited parent education programs designed to help children diagnosed with ADHD and disruptive behaviors can be helpful to families that may not be able to participate in "traditional" forms of mental health care. In short, the researchers want to know if a new program is acceptable and helpful for parents or caregivers looking for ways to help their child with problem behaviors related to ADHD. The researchers hope to enroll 60 families in the study. Half will be randomly assigned to participate in a 7-session therapy program and the other half will be asked to wait 24 weeks before being offered the treatment. Parents in the study will fill out questionnaires at week 1, week 14, and week 24.

The researchers' goal is to answer 2 specific questions. 1) Is this protocol acceptable to families and do they choose to participate and 2) Are the researchers able to accurately measure our outcomes of interest, specifically, changes in children's behavior problems, changes in parenting practices, and parents' perceptions of mental health care.

This study is focused on whether the intervention and study methods are acceptable. The researchers will compare the two groups to see if there are differences, but it would require a larger group of children and parents before the researchers can determine whether these differences are meaningful .

ELIGIBILITY:
Inclusion Criteria:

1. Children between ages 3-8 receiving services at the developmental pediatrics clinic at DH Lebanon referred by their physician for help with disruptive behaviors.
2. A diagnosis ADHD, ODD, Adjustment Disorder with Conduct, or Disruptive Behavior Disorder documented in the chart.
3. Family participating is capable of receiving in-person or telehealth care and treatment materials in English

Exclusion Criteria:

1. Primary concern that would indicate that behavioral parent training would not be the treatment of choice at the time of referral, including Autism Spectrum Disorder, previously untreated Post Traumatic Stress Disorder, OCD, or Reactive Attachment Disorder. The study clinician may also use clinical judgment that the intervention is inappropriate for a particular child's needs at any point during intervention.
2. Currently receiving outpatient therapy at the time of referral. The study will not exclude children on psychotropic medications, but will document medication status and changes to medication throughout treatment.
3. Severe history of physical or mental impairment (e.g., intellectual disability, global developmental delay). Child must be capable of verbal communication with a parent.
4. Children who are in foster care or are currently wards of the state.
5. Primary caregivers under 18 years of age.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in ADHD-5 | Measured at baseline, 14 weeks post baseline, and 24 weeks post baseline.
  This is a commonly used scale of inattention and hyperactivity with established norms by age group. The ADHD-5 has two sub-scales, Inattention and Hyperactivity, both comprised of 9 symptom-specific items that parents rate on a 4 point scale (0 = rarely to 4 = Very often) with higher numbers meaning more severe ADHD symptoms. Both scales also contain 6 items related to impairment in key areas of children's lives (exp: performance academically in school). Each impairment item is rated on a 4-point scale (0 = No Problem to 3 = Severe Problem) with higher numbers indicating greater impairment.
Change in Eyberg Child Behavior Inventory | Measured at baseline, 14 weeks post baseline, and 24 weeks post baseline.
  This is a commonly used scale to assess both the frequency of children's disruptive behaviors and the extent to which the parent finds the behaviors problematic. This measure is commonly used in the target age group to assess changes in symptoms during treatment. The Eyberg Child Behavior Inventory questionnaire is measured on two subscales for a series of phrases that describe a children's behavior. The first subscale is for indicating the frequency of the behavior using a scale of 1= never to 7 = Always; the second subscale indicates yes = 1 or no = 0 for whether the behavior is currently a problem for them. Reponses are totaled with a higher score indicating greater severity of child's behavior.
Change in Impairment Rating Scale | Measured at baseline, 14 weeks post baseline, and 24 weeks post baseline.
  This measure assesses the degree to which ADHD symptoms impair functioning. This is an analog scale that asks parents to go through each area of functioning in their child's life (social, academic, etc.) provide a short narrative about the problem their child faces and rate their level of impairment by marking a point on a line that can be divided into 100 segments. At one end of the spectrum is the anchor, "No Problem. Definitely does not need treatment or special services" and at the other end is the anchor "Extreme Problem. Definitely needs treatment or special services". Each item gets a score of 0-100 with higher scores indicating greater impairment.
Treatment Acceptability as evidenced by The Treatment Evaluation Inventory-Short Form | Measured only at 14 weeks after baseline in the treatment group.
  The Treatment Evaluation Inventory (TEI-SF) measure of treatment acceptability was specifically developed to evaluate parent trainings. It is a well-established quantitative measure of acceptance with an established cut-off score for 'moderate' acceptability. The TEI-SF is a single factor 9-item measure. Participants rate items on a 5-point scale 1 = Strongly Disagree to 5 = Strongly agree with one item reverse coded. Higher scores on the measure indicate higher treatment acceptability and a total score over 27 indicates moderate acceptability.
Treatment acceptability as evidenced by Parent Consumer Satisfaction Questionnaire | Measured only at 14 weeks after baseline in the treatment group.
  This measure of treatment acceptability was specifically developed to evaluate caregiver's perceptions of specific aspects of our parent training program. This measure assesses the 1) difficulty and 2) usefulness of each component of treatment. For each session activity (e.g., practice of skills with interventionist), parents rated if they found the activity useful and whether they found the activity difficult on a 7-point scale (1 = "Extremely Difficult/Extremely not useful" to 7 "Extremely Easy/Extremely Useful"). Parents used the same scale to rate each of the parenting skills they were taught during the program (e.g., praise, time-out). For this measure, higher numbers indicate that a skill was perceived positively (as useful and easy to implement) and lower numbers indicate difficulty and lower usefulness.
Changes in Clinician Global Impairment | Measured at baseline and 14 weeks after baseline. Treatment group only.
  This is a two item impairment scale used by the clinician to rate the impairment of the child before and after treatment. The two items are Severity of Illness and Global Improvement. Items are rated on a 7-point scale (1 = normal not at all/very much improved to 7 = Among the most extremely ill patients/very much worse). For this scale lower scores indicate better functioning and greater improvement.

SECONDARY OUTCOMES:
Changes in the Barriers to Children's Mental Health Survey | Measured at baseline and 14 weeks after baseline.
  We modified this measure from its original version to include a few additional items related to barriers to care. The original measure was developed to assess parental attitudes and beliefs about both the appropriateness of mental health care and the degree to which barriers including cost, travel, and other parent responsibilities might deter or facilitate the family's ability to participate in mental health treatment. The measure is divided into two parts: tangible barriers to care (e.g., missed time from work) and intangible barriers (being embarrassed if friends or family learned they were seeking help). There are 12 items on each sub-scale. Each item is rated on a 6-point scale with 1= "not a problem/strongly disagree" to 6 "a major problem/strongly agree". Several items are reverse coded and a single score is created for each domain. Higher scores on the measure indicate experiencing more severe barriers to care.
Changes in the Parenting Scale (PS; Rhodes & Leary, 2007). | Measured at baseline and 14 weeks after baseline.
  The parenting scale is a well validated and frequently used measure that assesses parents on three dimensions of negative-positive parenting 1) laxness, 2) verbosity, and 3) over reactivity. Each of the 30 items is rated on a 7-point scale. Each item provides two unique anchors at the ends of the scale that represent extremes of a parenting style. For example, on the laxness scale an items states "When my child misbehaves I..." The first anchor is "do something right away" and the anchor on the other end of the spectrum is "I do something later". Each item loads on one of the three factors with higher scores indicating more negative parenting styles.
Changes in Family Empowerment Scale | Measured at baseline and 14 weeks after baseline.
  The FES is commonly used with parents of children with many types of medical and psychiatric concerns and is used to assess how efficacious caregivers feel in their ability to help their child manage and concern and advocate for their child to receive appropriate care from others (e.g., doctors and school professionals). The scale has three factors related to empowerment: Family, Service Systems, and Community/Political. Each item is rated on 5-point scale (1= not true at all to 5 = very true). Higher scores indicate a greater sense of caregiver empowerment.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No